CLINICAL TRIAL: NCT00098267
Title: Collection of Dental Plaque and Saliva for Studies of Oral Microbial Colonization
Brief Title: Collection of Dental Plaque and Saliva for Studies of Bacterial Colonization of Teeth
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050051; 05-D-0051
Record Dates: First submitted 2006-07-12; First posted 2004-12-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-03

CONDITIONS: Healthy
Keywords: Bacteria; Biofilm Formation; Secretory Antibodies; Teeth; Health and Disease
MeSH Terms: conditions — Disease

SUMMARY:
This study will explore how bacteria colonize human teeth and how this process changes over the lifetime of individuals. It will include an investigation of transmission of bacteria that initiate colonization between adults and from adults to infants.

Selected NIH scientists and members of their immediate families, including infants, are eligible for this study. Participants provide a small sample of saliva and a sample of bacteria collected by rubbing a cotton swab over the surfaces of the lower four incisors. Adults collect and submit their own specimens; a dentist collects specimens from children.

DETAILED DESCRIPTION:
Interactions between different bacteria play an important role in biofilm development during primary colonization of the human tooth surface. Well studied examples of such interactions include the receptor polysaccharide (RPS)-mediated interactions between viridans group streptococci and other oral bacteria including type 2 fimbriated Actinomyces naeslundii. Previous studies have resulted in the identification of different structural, antigenic and molecular types of RPS on the streptococci that initiate colonization of the tooth surface. This information provides the basis for the current protocol, which addresses a number of important questions involving the nature of the commensal relationship that exists between biofilm-forming bacteria and the host. For example: (1) How many types of RPS are produced by the resident flora of an individual at any one time? (2) Does the resident population of RPS-producing clones change over the lifetime of the host? (3) Do individuals produce secretory antibodies against bacterial RPS, and if so, does this drive a change in the antigenic type of RPS produced? (3) When and how do infants acquire RPS-producing bacteria, before or after tooth eruption? To address these questions, we wish to collect and analyze samples of early dental plaque from the members of individual families. The collection of such samples will be accomplished by gently rubbing exposed tooth surfaces with a sterile cotton swab. Adult volunteers will also be asked to provide small samples of saliva, which will be assayed for the presence of specific anti-RPS antibodies. The sampling procedures proposed in this protocol do not present any significant risk to either adult or infant volunteers. The information gained from these studies, although not directly beneficial to these individuals, is expected to provide important insights into the commensal relationship that exists between biofilm-forming bacteria and the host. This in turn will contribute to an improved understanding of variables associated with the maintenance of oral health and the initiation of disease.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA

This is a pilot study with no inclusion or exclusion criteria other than availability. Participants will include Dr. Yoshida, his wife and their infant son and members of Dr. Cisar's family including his wife and adult children. Other NIH scientists and their infant children will also be included. All participants will be asked to sign the appropriate consent / assent forms.

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-12-02; Primary Completion 2009-08-03 (Actual); Study Completion 2009-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cisar JO, Sandberg AL, Abeygunawardana C, Reddy GP, Bush CA. Lectin recognition of host-like saccharide motifs in streptococcal cell wall polysaccharides. Glycobiology. 1995 Oct;5(7):655-62. doi: 10.1093/glycob/5.7.655. PMID 8608267
- [Background] Takahashi Y, Sandberg AL, Ruhl S, Muller J, Cisar JO. A specific cell surface antigen of Streptococcus gordonii is associated with bacterial hemagglutination and adhesion to alpha2-3-linked sialic acid-containing receptors. Infect Immun. 1997 Dec;65(12):5042-51. doi: 10.1128/iai.65.12.5042-5051.1997. PMID 9393794
- [Background] Takahashi Y, Ruhl S, Yoon JW, Sandberg AL, Cisar JO. Adhesion of viridans group streptococci to sialic acid-, galactose- and N-acetylgalactosamine-containing receptors. Oral Microbiol Immunol. 2002 Aug;17(4):257-62. doi: 10.1034/j.1399-302x.2002.170409.x. PMID 12121477